CLINICAL TRIAL: NCT01888783
Title: Comparison of Two Measures of Tactile Acuity in CRPS Type I Patients , Patients With a Neuropathy of the Median Nerve and Healthy Controls.
Brief Title: Two Measures of Tactile Acuity in CRPS Type I Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Prof. Dr. med Christoph Maier, Head Dep. of Pain Medicine, Ruhr University of Bochum
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GOT_CRPS2013
Record Dates: First submitted 2013-06-25; First posted 2013-06-28 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-06

CONDITIONS: CRPS Type I of the Upper Extremity; Neuropathy of the Median Nerve; Healthy Controls
Keywords: CRPS Type I; tactile acuity; 2-point-discrimination; Grating Orientation Task; sensory signs
MeSH Terms: conditions — Reflex Sympathetic Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CRPS Type I (Experimental): Patients diagnosed with complex regional pain syndrome type I of the upper limb
  Interventions: Other: Tactile acuity measured by 2PD and the GOT
- Median Nerve Neuropathy (Active Comparator): Patients diagnosed with a neuropathy of the median nerve of the upper limb.
  Interventions: Other: Tactile acuity measured by 2PD and the GOT
- Healthy Controls (Active Comparator): Healthy adult persons.
  Interventions: Other: Tactile acuity measured by 2PD and the GOT

INTERVENTIONS:
Other: Tactile acuity measured by 2PD and the GOT — For a detailed description of the methods see "outcome measures"
  Other Names: 2-point-discrimination (2PD); Grating Orientation Task (GOT)

SUMMARY:
This study aims to investigate whether two different measures of tactile acuity lead to comparable results in patients diagnosed with CRPS Type I of the upper extremity. Additionally patients with a neuropathy of the median nerve and healthy controls are included.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CRPS Type I according to the "Budapest Criteria"
* Patients diagnosed with a neuropathy of the median nerve
* Healthy Controls,matched in age and gender to both patient cohorts

Exclusion Criteria:

* intolerable hyperalgesia
* lesions at the fingertips
* high grade digit contracture
* central neurologic disorders
* psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
tactile acuity as measured by 2-point-discrimination | unique measurement of maximal one hour duration
  Thresholds on the tip of the index finger of boths hands are assessed using the method of constant stimuli. One single needle and seven pairs of needles with different spacings are tested in randomized order. After each presentation, the subject has to report the sensation of one or two needles by answering immediately "one" or "two." Each distance is presented eight times resulting in 64 single decisions. The summed responses are plotted against distance as a psychometric function for absolute threshold and get fitted by a binary logistic regression. Thresholds are taken from the fit at the distance at which 50% correct answers are given
tactile acuity as measured by the Grating Orientation Task (GOT) | unique measurement of maximal half an hour duration
  Stimuli are taken from a set of dome-shaped plastic gratings with equal groove and ridge widths. Gratings are applied to the immobilized distal fingerpad of the index finger of boths hand with the ridges oriented either along or across the long axis of the finger in randomized sequences of the two alternatives. Subjects have to report the orientation of the gratings as "along" or "across". The largest groove widths in the set is 6mm, the minimal width is 0.5mm. Thresholds were taken from the groove width at which the performance was 75% correct. Unless the performance is exactly 75% for a particular grating, interpolation between gratings spanning the 75% correct responses ared used

OTHER OUTCOMES:
Touch threshold for light touch | unique measurement, duration approx. 5 minutes
  Touch thresholds are taken from a set of von Frey filaments (0.25 mN - 512 mN). Touch sensitivity is investigated by using a staircase procedure during which subjects are required to close their eyes and report when they perceive an indentation of the skin on the fingerpad of the index finger. The applied forces are decreased in a stepwise manner until the subject no longer perceives the stimulus (lower boundary) and then increased until the stimulus is perceived again (upper boundary). This procedure is repeated 5 times resulting in 10 values that are averaged to provide the touch threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Maier, Prof. Dr., Study Chair — Ruhr University Bochum
Locations (1):
- Department of Pain Medicine, BG Universitätsklinikum Bergmannsheil GmbH, Bochum, Germany